CLINICAL TRIAL: NCT01622140
Title: Prospective Comparison of the Tuberculin Skin Test and Interferon-Gamma Release Assays in Diagnosing Infection With Mycobacterium Tuberculosis and in Predicting Progression to Tuberculosis
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CDC-TBESC-TO1
Record Dates: First submitted 2012-06-04; First posted 2012-06-18 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Latent Tuberculosis Infection; Tuberculosis
Keywords: T-SPOT.TB; QuantiFERON-TB Gold In-Tube; Latent tuberculosis infection; Tuberculin skin test; Discordance; Predictive value; Tuberculosis disease development
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective cohort study of persons tested for latent tuberculosis infection at either high risk for exposure to Mycobacterium tuberculosis or high risk for progression to tuberculosis disease. The study will assess the relative performance and cost of three diagnostic tests for latent tuberculosis infection (tuberculin skin test, QuantiFERON-TB Gold In-Tube, and T-SPOT.TB) and will examine the rates of positive results among the cohort. This study will also determine the risk and rate of progression to active TB disease, overall and by the results of the three tests.

ELIGIBILITY:
1. Study participants must be at high risk for latent tuberculosis infection or at high risk for progression to tuberculosis disease, including being a:

   • Close contact of a person with pulmonary tuberculosis who is part of a current contact investigation and the index/source case meets the following criteria:
   1. Culture-positive, OR
   2. Culture-negative and smear positive and nucleic acid amplification test-positive.

   Participants may be enrolled before the culture results for the index/source case are available. If the criteria described above are not met once results are available, the participant will be terminated from the study and any collected data will be immediately destroyed.

   A close contact is defined as spending 15 or more hours over a week's period in a shared airspace with a person with active pulmonary tuberculosis while that person was presumed to be infectious.
   * Foreign-born person from a high risk country.
   * Foreign-born person from a medium risk country who moved to the United States within the past 5 years.
   * Person who has spent at least 30 days in total in a high risk country within the last 5 years.
   * Person belonging to a population with a prevalence of latent tuberculosis infection ≥ 25% as demonstrated by local surveys. These populations will vary by site; examples include Mexican immigrants in San Diego, California or homeless drug users in Baltimore, Maryland.
   * HIV-positive person.
2. Study participants (or a parent/guardian, if applicable) must be willing and able to provide informed consent.

4.2 Subject Exclusion Criteria

Subjects meeting any of the exclusion criteria will be excluded from study enrollment.

1. People with known current active tuberculosis.
2. People with a previous anaphylactic reaction to tuberculin.
3. Persons currently being treated for latent tuberculosis infection.
4. Persons anticipating or scheduled to permanently leave the United States (e.g., tourists, visiting scholars, exchange students) in less than 2 years from the time of proposed study enrollment.
5. Foster children.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals at high risk for latent tuberculosis infection or at high risk for progression to tuberculosis from health clinics, hospitals, or health departments at the 10 Tuberculosis Epidemiologic Studies Consortium sites within the United States: California Department of Public Health, Denver Health and Hospital Authority, Duke University, Emory University, Hawaii Department of Health, Maricopa County Department of Public Health, Maryland Department of Public Health, Public Health Seattle-King County, University of Florida Board of Trustees, and University of North Texas Health Science Center
Sampling Method: Non-Probability Sample
Enrollment: 21334 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Latent tuberculosis infection | 3 days
Tuberculosis disease at 6 months | 6 months
Tuberculosis disease at 12 months | 12 months
Tuberculosis disease at 18 months | 18 months
Tuberculosis disease at 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ho, MD, Principal Investigator — Centers for Disease Control and Prevention; Dolly Katz, PhD, Principal Investigator — Centers for Disease Control and Prevention; Thara Venkatappa, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (10):
- United States (10):
  - Maricopa County Department of Public Health, Phoenix, Arizona
  - California Department of Public Health, Richmond, California
  - Denver Health and Hospitals Authority, Denver, Colorado
  - University of Florida Board of Trustees, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Hawaii Department of Health, Honolulu, Hawaii
  - Maryland Department of Public Health, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Public Health Seattle-King County, Seattle, Washington

REFERENCES:
- [Derived] Ayers T, Hill AN, Raykin J, Mohanty S, Belknap RW, Brostrom R, Khurana R, Lauzardo M, Miller TL, Narita M, Pettit AC, Pyan A, Salcedo KL, Polony A, Flood J; CDC Tuberculosis Epidemiologic Studies Consortium. Comparison of Tuberculin Skin Testing and Interferon-gamma Release Assays in Predicting Tuberculosis Disease. JAMA Netw Open. 2024 Apr 1;7(4):e244769. doi: 10.1001/jamanetworkopen.2024.4769. PMID 38568690
- [Derived] Ho CS, Feng PI, Narita M, Stout JE, Chen M, Pascopella L, Garfein R, Reves R, Katz DJ; Tuberculosis Epidemiologic Studies Consortium. Comparison of three tests for latent tuberculosis infection in high-risk people in the USA: an observational cohort study. Lancet Infect Dis. 2022 Jan;22(1):85-96. doi: 10.1016/S1473-3099(21)00145-6. Epub 2021 Sep 6. PMID 34499863
- [Derived] Ahmed A, Feng PI, Gaensbauer JT, Reves RR, Khurana R, Salcedo K, Punnoose R, Katz DJ; TUBERCULOSIS EPIDEMIOLOGIC STUDIES CONSORTIUM. Interferon-gamma Release Assays in Children <15 Years of Age. Pediatrics. 2020 Jan;145(1):e20191930. doi: 10.1542/peds.2019-1930. PMID 31892518
- [Derived] Stout JE, Wu Y, Ho CS, Pettit AC, Feng PJ, Katz DJ, Ghosh S, Venkatappa T, Luo R; Tuberculosis Epidemiologic Studies Consortium. Evaluating latent tuberculosis infection diagnostics using latent class analysis. Thorax. 2018 Nov;73(11):1062-1070. doi: 10.1136/thoraxjnl-2018-211715. Epub 2018 Jul 7. PMID 29982223